CLINICAL TRIAL: NCT06483347
Title: Intra-tumor Delivery of Double Checkpoint Inhibitors, Chemodrug, and/or Bevacizumab Therapy as First Line for Inoperable Lung Cancer
Brief Title: Checkpoint Inhibitor Combinations Therapy as First Line for Inoperable Lung Cancer Via IT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZ-IT-ICI-LC 1line-025
Record Dates: First submitted 2024-06-23; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Inoperable Disease
Keywords: Inoperable lung cancer; Intra-tumor injection; Immunotherapy; First line therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Idarubicin; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- IT injection of double ICI (Experimental): Arm 1: intra-tumor injection of double ICIs only.
  Interventions: Drug: ipilimumab+pembrolizumab or ipilimumab+durvalumab, idarubicin, bevacizumab
- IT injection of double ICI and chemodrug (Experimental): Arm 2: intra-tumor injection of double ICIs and a chemodrug.
  Interventions: Drug: ipilimumab+pembrolizumab or ipilimumab+durvalumab, idarubicin, bevacizumab
- IT injection of double ICI and chemodrug plus bevacizumab (Experimental): Arm 3: intra-tumor injection of double ICIs, a chemodrug, and bevacizumab.
  Interventions: Drug: ipilimumab+pembrolizumab or ipilimumab+durvalumab, idarubicin, bevacizumab

INTERVENTIONS:
Drug: ipilimumab+pembrolizumab or ipilimumab+durvalumab, idarubicin, bevacizumab — This study has 3 subgroups:
  Arm 1. Ipilimumab +pembrolizumab or Ipilimumab +durvalumab is administrated with a total dose of 1-2mg/kg via intra-tumor fine needle injection in 10 min, every 3 weeks.
  Arm 2. Ipilimumab +pembrolizumab or Ipilimumab +durvalumab combined with idarubicin is administrated via intra-tumor fine needle injection in 15 min, every 3 weeks.
  Arm 3. Ipilimumab +pembrolizumab or Ipilimumab +durvalumab combined with idarubicin plus bevacizumab is administrated via intra-tumor fine needle injection in 20 min, every 3 weeks.
  Other Names: Local ICIs.

SUMMARY:
This trial is designed to investigate the safety, response rates and survival outcomes of patients with inoperable lung cancer by infusion of CTLA4, PD1 and PDL1 antibodies combination with chemodrug or/and bevacizumab through intra-tumor (IT).

DETAILED DESCRIPTION:
Antibodies against CTLA4, PD1 and PDL1 are representative drugs for the check-points inhibitory agents, and their clinical indications have been approved in various types of tumors, including advanced melanoma, non-small cell lung cancer, renal cell carcinoma, and classical Hodgkin's lymphoma and late recurrent head and neck squamous cell carcinoma patients, et al. Those drugs are regularly systemically administrated by vein infusion, however, local delivery of those drugs via interventional radiology technique including trans-artery or intra-tumor injection may increase the local drug concentration of the tumor, improve the efficacy, and reduce systemic adverse reactions. CTLA4 antibody ipilimumab has been widely effectively using to combine with PD1 or PDL1 antibody and this study is to combine ipilimumab and PD1 antibody or PDL1 antibody, so called double checkpoint inhibitors combination therapy, as first line for inoperable lung cancer via intra-tumor admistration. To the investigator's knowledge, no studies have been developed on the safety, efficacy and survival benefit of the double checkpoint inhibitors combination therapy for cancer patients as first line via intra-tumor delivery.

This phase II clinical trial is designed to assess the safety and survival benefit of ipilimumab and pembrolizumab or durvalumab combination with or without chemodrug or bevacizumab as first line therapy on patients with inoperable lung cancer, including PFS, ORR, DCR, and median survival time.

ELIGIBILITY:
Inclusion Criteria:

1. Cytohistological confirmation is required for diagnosis of cancer.
2. Signed informed consent before recruiting.
3. Age above 18 years with estimated survival over 3 months.
4. Child-Pugh class A or B/Child score > 7; ECOG score < 2
5. Tolerable coagulation function or reversible coagulation disorders
6. Laboratory examination test within 7 days prior to procedure: WBC≥3.0×10E9/L; Hb≥90g/L； PLT ≥50×10E9/L；INR < 2.3 or PT < 6 seconds above control；Cr ≤ 145.5 umul/L；Albumin > 28 g/L；Total bilirubin < 51 μmol/L
7. At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1.
8. Birth control.
9. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

1. Patients participated in clinical trials of equipment or drugs (signed informed consent) within 4 weeks;
2. Patients accompany by ascites, hepatic encephalopathy and esophageal and gastric varices bleeding;
3. Any serious accompanying disease, which is expected to have an unknown, impact on the prognosis, include heart disease, inadequately controlled diabetes and psychiatric disorders;
4. Patients accompanied with other tumors or past medical history of malignancy;
5. Pregnant or lactating patients, all patients participating in this trial must adopt appropriate birth control measures during treatment;
6. Patients have poor compliance.

   Any contraindications for hepatic arterial infusion procedure:

   A.Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 50%).

   B.Renal failure / insufficiency requiring hemo-or peritoneal dialysis. C.Known severe atheromatosis. D.Known uncontrolled blood hypertension (> 160/100 mm/Hg).
7. Allergic to contrast agent;
8. Any agents which could affect the absorption or pharmacokinetics of the study drugs
9. Other conditions that investigator decides not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety of IT delivery of drugs combination treatment | 5 years
  Safety will be assessed by recording all types of advise effects upon and after the treatment.
Progression-free survival | 5 years
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per RECIST 1.1) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment.
Disease control rate | 5 years
  Disease control rate will be defined as objective response rate + steady disease rate.
Duration of remission (DOR) | 5 years
  DOR will be defined as the duration of the cancer remission.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival (OS) will be defined as the elapsed time from the enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will occur every 12 weeks (±1 month) until death or withdrawal of consent from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China